CLINICAL TRIAL: NCT05926011
Title: Efficacy of RGn600 in Patients With Mild-to-moderate Alzheimer's Disease: a Pivotal, Sham-controlled, Randomized, Double-blind, Multicentric Investigation (LIGHT4LIFE)
Brief Title: Efficacy of RGn600 in Patients With Mild-to-moderate Alzheimer's Disease
Acronym: LIGHT4LIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: REGEnLIFE SAS (Industry)
Collaborators: RCTs (Industry); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIGHT4LIFE; 2022-A02556-37 (Registry Identifier: IDRCB number. French competent authority : Agence Nationale de sécurité du médicament et des produits de santé (ANSM))
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; Neurostimulation; Optics and photonics; Photobiomodulation; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Medical Device
MeSH Terms: conditions — Alzheimer Disease; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: An interventional, prospective, multicentric, randomized, comparative and double-blinded pivotal clinical investigation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active RGn600 (Experimental): RGn600 with a 10 Hz-pulsed wave mode light emission
  Interventions: Device: RGn600
- Sham (Sham Comparator): Inactivated RGn600
  Interventions: Device: RGn600 Sham

INTERVENTIONS:
Device: RGn600 — RGn600 with a 10 Hz-pulsed wave mode light emission
  Arms: Active RGn600
Device: RGn600 Sham — RGn600 inactivated
  Arms: Sham

SUMMARY:
This is a controlled investigation, with randomization of the patients, which aims at demonstrating the efficacy of device RGn600 in treating patients with mild-to-moderate Alzheimer's disease (AD). RGn600 is a non-invasive medical device which is applied on the head (helmet) and on the abdomen (abdominal belt). It combines 2 technologies:

* PhotoBioModulation (PBM), which involves exposure to light from the red to near-infrared wavelengths using lasers and Light Emitting Diodes (LEDs)
* Static Magnetic Stimulation (SMS), which consists in the application of a static magnetic field.

Considering previous investigations, this innovative technology could reduce inflammation on the brain-gut axis, implicated in the development of Alzheimer's disease.

DETAILED DESCRIPTION:
This multicentric investigation is planned to include 108 patients in France who will be followed up to 52 weeks.

Patients meeting all eligibility criteria will be randomized on a 1: 1 ratio into one of the two following treatment groups: active RGn600 device or sham device (inactivated RGn600). The site investigation teams and patients/caregivers will be blinded. The device will be applied to the patients during 26 weeks through 20-min onsite sessions following the below pattern:

* 5 treatment sessions per week from Week 1 (W1) to W8
* 3 treatment sessions per week from W9 to W16
* 2 treatment sessions per week from W17 to W26 Throughout the investigation, patients will be treated per randomization with the device initially allocated by the IWRS.

Follow-up will continue up to W52 ± 2 weeks

At inclusion visit, after verification of the eligibility criteria, data regarding patients will be collected: demographic data, date of AD diagnosis, comorbidities, concomitant medications, sociological data. A blood sample for APOE genotyping will be also performed.

Endpoints will be evaluated during 4 onsite visits at Day 0 (Inclusion, randomization to the active or sham group and first treatment session), W8 (last treatment session of), W26 (last treatment session of) and W52 ± 2 weeks. During these visits:

* Patient's cognition and autonomy will be assessed through neurological scales and/or neuropsychological tests
* Patient's quality of life and medico-economic interest of RGn600 treatment with regards to healthcare consumption will be assessed through questionnaires fulfilled by the patient himself/herself with the help of his/her caregiver
* The safety of RGn600 will be assessed : collection of all AEs and device deficiencies, blood samples for safety analysis, clinical exams

Within the context of this investigation, a biobank will be created based on blood, fecal and saliva samples of patients included by Toulouse University Hospital Gerontopole site:

* Blood samples will be collected for all patients included by this site (at D0, W26 and W52)
* Fecal samples will be collected for the first 30 consecutive patients included by this site (at D0, W26 and W52).
* Saliva samples will be collected for the patients included by this site after the substantial modification approval (at D0, W26 and W52).

The biobank will be located at the site. The objective of this biobank will be to perform subsequent analysis on blood samples of AD blood markers. Other analyses might be conducted on blood, fecal and saliva samples as well such as Inflammatory blood markers (iAGE), fecal microbiota and metabolome and salivary micro RiboNucleic Acid (microRNAs)

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 55 to 85 years old (both included)
* Diagnosed with AD according to McKhann et al. international criteria dated 2011
* With mild-to-moderate AD, i.e., 10 ≤ MMSE score ≤ 26
* With blood analyses results (for: thyroid-stimulating hormone, vitamin B12, folate, complete blood count including platelets, electrolytes including calcium, creatinine, clearance, alanine aminotransferase, aspartate aminotransferase, bilirubin, coagulation, C-reactive protein) dated less than 1 year ago in line with AD diagnosis, as deemed by the investigator
* With brain Computed Tomography (CT) or/and Magnetic Resonance Imaging (MRI) scan dated less than 1 year ago in line with AD diagnosis, as deemed by the investigator
* In case of treatment with AD symptomatic treatments (memantine and acetylcholinesterase inhibitors) and psychotropic treatments (anxiolytics, antidepressants and neuroleptics): with a stable dose of such treatments 4 weeks before inclusion
* Who has a caregiver who is sufficiently and regularly present and can help the patient throughout the investigation, as deemed by the investigator
* Affiliated to French social security
* Who provided, with his/her caregiver, a dated and signed informed consent form.

Exclusion Criteria:

* Patient protected by a French legal measure ("sauvegarde de justice", "tutelle" or "curatelle")
* Patient deprived of liberty or hospitalized without consent
* Non-menopausal woman
* Patient taking a disease-modifying treatment such as the Leqembi® or any other disease-modifying treatment that may be authorized in France before the end of the study
* Patient living in a medical facility
* Patient who experienced a surgery at the treatment application area (abdomen or head) within 3 months prior inclusion
* Patient with skin lesions on the treatment application area (abdomen or head)
* Patient with a short-term life-threatening pathology (e.g., evolving cancer; non-stable heart failure; severe hepatic, renal or respiratory failure, etc.)
* Patient diagnosed with a stroke within 3 months prior inclusion
* Patients with ferromagnetic material (i.e., iron, nickel, cobalt or any metal alloy) on or near the head or abdomen, or implanted with a pacemaker
* Patient with a risk of epileptic seizure
* Patient with a genetic form of AD
* Patient with major physical or neurosensorial disorders that may interfere with neurological assessments
* Patient with chronic psychosis or psychotic episodes
* Patient addicted to alcohol or drugs
* Patient with known and non-supplemented vitamin B12 and folic acid deficiencies
* Patient with known untreated hypothyroidism
* Patient who participated to another investigation/study involving the use of an investigational medical device/drug within the 30 days prior inclusion
* Patient not able to meet treatment sessions as deemed by the investigator
* Patient not able to complete requested investigation assessments as deemed by the investigator.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evolution of patient's cognition between Day 0 and Week 26 as measured with the AD Assessment Scale-cognitive subscale (ADAS-cog) score | Day 0, Week 26
  Absolute change (Week 26-Day 0) in ADAS-cog score

SECONDARY OUTCOMES:
Evolution of patient's cognition from Day 0 to Week 8, from Day 0 to Week 52 and from Week 26 to Week 52 as measured with the AD Assessment Scale-cognitive subscale (ADAS-cog) score | Day 0, Week 8, Week 26, Week 52
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's cognitive functions | Day 0, Week 26, Week 52
  Evolution of the score of the Mini Mental State Examination (MMSE)
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's cognitive functions | Day 0, Week 26, Week 52
  Evolution of the score of the Category Naming Test (CNT)
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's cognitive functions | Day 0, Week 26, Week 52
  Evolution of the scores of the Digit Symbol Substitution Test (DSST)
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's cognitive functions | Day 0, Week 26, Week 52
  Evolution of the score of the Trail Making Test part A and B (TMT A & B)
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's cognitive functions | Day 0, Week 26, Week 52
  Evolution of the score of the Clinical Dementia Rating - Sum of Boxes (CDR-SB) scale
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's cognitive functions | Day 0, Week 26, Week 52
  Evolution of the score of the AD Composite Score (ADCOMS)
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's cognitive functions | Day 0, Week 26, Week 52
  Evolution of the score of the Digit span test
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's autonomy | Day 0, Week 26, Week 52
  Evolution of the Instrumental Activities of Daily Living (IADL) questionnaire score
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's Overall clinical response | Day 0, Week 26, Week 52
  Evolution of the Clinical Global Impression (CGI) scale score
Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's Quality of life | Day 0, Week 26, Week 52
  Evolution of the EuroQoL 5 Dimensions-5 Levels (EQ-5D-5L) score
Incidence of Adverse Events (AEs) | Throughout the investigation (from Day 0 to Week 52)
  Proportion of subjects with at least one Adverse Event (AE)
Incidence of RGn600's Adverse Device Effects (ADEs) | Throughout the investigation (from Day 0 to Week 52)
  Proportion of subjects with at least one Adverse Device Effect (ADE)
Incidence of RGn600's Device Deficiencies (DDs) | Throughout the investigation (from Day 0 to Week 52)
  Proportion of subjects with at least one Device Deficiency (DD)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of Complete blood count, including platelets
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of electrolytes, including calcium
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of Creatinine
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of creatinine clearance
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of urea
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of ASpartate AminoTransferase (ASAT)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of ALanine AminoTransferase (ALAT)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of Gamma-GT
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of ALkalyne Phosphatase (ALP)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of level of safety blood markers | Day 0, Week 8, Week 26, Week 52
  Change from baseline (Day 0) of level of bilirubin
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of Blood pressure | Day 0, Week 8, Week 26, Week 52
  Measure of Blood pressure (mmHg)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of Weight | Day 0, Week 8, Week 26, Week 52
  Measure of Weight (Kg)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of Heart rate | Day 0, Week 8, Week 26, Week 52
  Measure of Heart rate (beats/min)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of Temperature | Day 0, Week 8, Week 26, Week 52
  Measure of Temperature (°C)
Evolution from Day 0 to Week 8, Day 0 to Week 26 and from Day 0 to Week 52 of ElectroCardioGram (ECG) interpretation | Day 0, Week 8, Week 26, Week 52
  ElectroCardioGram (ECG) interpretation (Normal / Abnormal - Abnormality description)
Medico-economic interest of RGn600 treatment with regards to healthcare consumption | Day 0, Week 26
  Resource Utilization in Dementia (RUD) questionnaire filled in by the patient/caregiver.

OTHER OUTCOMES:
[Exploratory endpoint from biobanking] Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's AD blood markers | Day 0, Week 26, Week 52
  Evolution of Aβ42/Aβ40 ratio
[Exploratory endpoint from biobanking] Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's AD blood markers | Day 0, Week 26, Week 52
  Evolution of level of Glial Fibrillary Acidic Protein (GFAP)
[Exploratory endpoint from biobanking] Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's AD blood markers | Day 0, Week 26, Week 52
  Evolution of level of NeuroFilament Light (NFL) protein
[Exploratory endpoint from biobanking] Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's AD blood markers | Day 0, Week 26, Week 52
  Evolution of level of Phosphorylated tau 217 (p-tau 217)
[Exploratory endpoint from biobanking] Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's microbiota | Day 0, Week 26, Week 52
  Evolution of microbiota
[Exploratory endpoint from biobanking] Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's metabolome | Day 0, Week 26, Week 52
  Evolution of metabolome
[Exploratory endpoint from biobanking] Evolution from Day 0 to Week 26 and from Day 0 to Week 52 of patient's AD saliva markers | Day 0, Week 26, Week 52
  Evolution of microRNAs

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BLIVET, Study Director — REGEnLIFE SAS; Jacques TOUCHON, Study Chair — Montpellier University; Julien DELRIEU, Principal Investigator — Toulouse University Hospital Gerontopole
Locations (6):
- France (6):
  - CHIC Castres Mazamet Site Autan, Castres
  - CH Lavaur, Lavaur
  - Hôpital Lariboisière, Paris
  - Hôpital Broca, Paris
  - Hôpital de la Timone,, Timone
  - Toulouse University Hospital Gerontopole, Toulouse

IPD SHARING:
Plan to Share IPD: No